CLINICAL TRIAL: NCT06018558
Title: A Phase 1/2 Study to Assess the Safety And Efficacy Of OCU410 For Geographic Atrophy Secondary To Dry Age-Related Macular Degeneration
Brief Title: Study to Assess the Safety and Efficacy of OCU410 for Geographic Atrophy
Acronym: ArMaDa
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ocugen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: OCU410-101
Record Dates: First submitted 2023-06-30; First posted 2023-08-30 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Intervention Model Description: Study will be conducted in 2 phases:
  Phase 1 will be 3+3 design will be used for sequential dose-escalation cohorts in which subjects will receive a single subretinal injection of OCU410 in the study eye.
  Phase 2 is a dose-expansion phase of the study, where up to 51 subjects will be randomized in 1:1:1 ratio to either two OCU410 dose groups (n=17 per group) or to an untreated control group (n=17).
Who Masked: Outcomes Assessor
Masking Description: The following team members will be masked:
  Bio-Statistician, Data Programmer, Imaging Reading Center Team, Head of Clinical Development and Medical Affairs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase1 Dose Escalation- Low Dose (2.5×10E10 vg/mL): (Experimental): Low Dose (2.5×10E10 vg/mL): Subjects will receive a subretinal injection of OCU410 in the low dose concentration.
  Interventions: Genetic: OCU410
- Phase1 Dose Escalation- Medium Dose (5×10E10 vg/mL): (Experimental): Medium Dose (5×10E10 vg/mL): Subjects will receive a subretinal injection of OCU410 in the medium dose concentration.
  Interventions: Genetic: OCU410
- Phase1 Dose Escalation- High Dose (1.5×10E11 vg/mL): (Experimental): High Dose (1.5×10E11 vg/mL): Subjects will receive a subretinal injection in the high dose concentration.
  Interventions: Genetic: OCU410
- Phase 2 Dose Expansion: Maximum tolerated dose (MTD) from Phase 1-Randomized Arm (Experimental): Maximum tolerated dose (MTD) from Phase 1: Subjects will receive a subretinal injection in the MTD concentration.
  Interventions: Genetic: OCU410
- Phase 2 Dose Expansion: Lower Dose from Phase 1-Randomized Arm (Experimental): Subjects will receive a subretinal injection of OCU410 in a Lower Dose concentration.
  Interventions: Genetic: OCU410
- Control Arm (No Intervention): No Intervention Control Arm: Subject will not receive any active study intervention

INTERVENTIONS:
Genetic: OCU410 — Subretinal administration of OCU410
  Arms: Phase 2 Dose Expansion: Lower Dose from Phase 1-Randomized Arm; Phase 2 Dose Expansion: Maximum tolerated dose (MTD) from Phase 1-Randomized Arm; Phase1 Dose Escalation- High Dose (1.5×10E11 vg/mL):; Phase1 Dose Escalation- Low Dose (2.5×10E10 vg/mL):; Phase1 Dose Escalation- Medium Dose (5×10E10 vg/mL):

SUMMARY:
This is a Phase 1/2 Study to Assess the Safety and Efficacy of OCU410 for Geographic Atrophy Secondary to Dry Age-Related Macular Degeneration (AMD).

This is a multicenter study, which will be conducted in two phases and will enroll up to a total of 60 subjects.

DETAILED DESCRIPTION:
Name of Sponsor/Company:

Ocugen, Inc. 11 Great Valley Parkway Malvern, PA 19355

Name of Investigational Product: OCU410

Name of Active Ingredient:

Adeno-associated viral vector 5 human RORA (AAV5-hRORA) Protocol Number: OCU410-101 Phase: 1/2 Country: US

Title of Study:

A Phase 1/2 Study to Assess the Safety and Efficacy of OCU410 for Geographic Atrophy Secondary to Dry Age-Related Macular Degeneration.

Study Center(s): Approximately 14 clinical study centers in the US.

Background:

Age-related Macular Degeneration (AMD) is an ocular disease where macular degenerative occurs. AMD manifests in two forms, Dry (nonexudative, atrophic) AMD and Wet (exudative, neovascular) AMD. Geographic atrophy (GA) is an advanced stage of dry AMD that affects nearly 1 million people in the US and 5 million people worldwide, with its prevalence increasing exponentially with age. It leads to progressive and irreversible loss of visual function due to the growth of atrophic lesions that destroy the retinal cells responsible for vision.

OCU410 Product Information:

Ocugen, Inc., has developed a proprietary modifier gene therapy platform, OCU410, as the second agent in a novel class of NHR-based gene modifier therapy for patients with dry AMD. The proposed indication for OCU410 (AAV5-hRORA) is for the treatment of GA secondary to dry AMD. The drug product is a sterile ophthalmic suspension for subretinal injection. OCU410 therapy regulates gene pathways contributing to GA by restoring homeostasis in the eye and thereby serving as a therapeutic candidate for dry AMD. The modifier gene therapy platform is a new way of addressing a genetic disease arising through a multitude of genetic mutations in various genes but leading to the same end result (phenotype) of a diseased condition.

This study will be conducted in two phases enrolling up to 60 subjects. Treated subjects will receive a single subretinal injection of OCU410 in the study eye.

Phase 1 is a multicenter, open-label, dose-ranging/dose-escalating study with a 3+3 design enrolling 9 subjects.

Phase 2 is a dose-expansion phase of the study, where up to 51 subjects will be randomized in 1:1:1 ratio to either two OCU410 dose groups (n=17 per group) or to an untreated control group (n=17).

.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 50 years of age or older.
2. BCVA of approximately 21 letters or more using Early Treatment Diabetic Retinopathy Study (ETDRS) chart (20/320 Snellen equivalent).
3. Fundus autofluorescence (FAF) imaging shows:

   1. Total GA area ≥2.0 and ≤20.5 mm2 (1 and 8 disk areas [DA], respectively)
   2. If GA is multifocal, at least one focal lesion must be ≥1.25 mm2 (0.5 DA), with the overall aggregate area of GA as specified above in 3.a
   3. The entire GA lesion must be completely visualized on the macula-centered image and must be able to be imaged in its entirety, and not contiguous with any areas of peripapillary atrophy
   4. Presence of any pattern of hyper-autofluorescence in the junctional zone of GA
4. Subjects who had prior treatment with an approved drug for AMD, e.g. Izerway® (Avacincaptad pegol) or Syfovre® (Pegcetacoplan injection) can be included, after a washout period of at least 3 months in study eye. Subjects can receive an approved drug for AMD in the fellow eye, if required.

Exclusion Criteria:

1. Previous treatment with a gene-therapy or cell therapy product
2. GA due to causes other than AMD such as Stargardt disease, cone rod dystrophy or toxic maculopathies like Plaquenil maculopathy. However, benign conditions of the vitreous or peripheral retina are not exclusionary (i.e., pavingstone degeneration).
3. Spherical equivalent of the refractive error demonstrating > 6 diopters of myopia or an axial length >26 mm, inability to fixate, uncontrolled glaucoma, advanced cataract, corneal abnormalities, medium haze, and other retinal pathologies.
4. Any history or current evidence of exudative ("wet") AMD including any evidence of retinal pigment epithelium rips, branch retinal artery or vein occlusion, corneal transplant, or evidence of neovascularization anywhere in the retina based on fluorescein angiogram.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2026-02-17 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Safety (Participants With Ocular and Non-ocular AEs (Adverse Events) and SAEs (Serious Adverse Events)) | 12 months (Screening to 12 months post OCU410 administration)
  The primary endpoint is safety, determined by the number of ocular and non-ocular Study Drug-related adverse events (SDAE), treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs).
Change in anatomy of ocular structures using Slit Lamp Biomicroscopy | 12 months (Screening to 12 months post OCU410 administration)
  We will use Slit-lamp Biomicroscopy to visualize the anatomy of ocular structures before and after sub-retinal injections and follow-up visits.
Change in anatomy of ocular structures using Indirect ophthalmoscopy | 12 months (Screening to 12 months post OCU410 administration)
  We will use Indirect ophthalmoscopy to visualize the anatomy of ocular structures before and after sub-retinal injections and follow-up visits.
Change from baseline in BCVA (Best Corrected Visual Acuity) | 12 months (Screening to 12 months post OCU410 administration)
  Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. A higher score represents better vision.
Change in Low Luminance Visual Acuity | 12 months (Screening to 12 months post OCU410 administration)
  Measured by letter score. A higher score represents better vision
Change in the Intraocular Pressure (mmHg) | 12 months (Screening to 12 months post OCU410 administration)
  Measured by applanation or rebound tonometry with confirmation with Goldmann tonometer if IOP is outside normal range (8-21mmHg).

SECONDARY OUTCOMES:
Humoral and cellular immune response | 12 months (Screening to 12 months post OCU410 administration)
  Blood samples will be collected for the assessment. The secondary safety endpoints include change from baseline in Humoral and cellular immune response in response to OCU410 administration
Shedding of viral vector | 12 months (Screening to 12 months post OCU410 administration)
  Blood samples will be collected for the assessment to determine AAV vector shedding in systemic circulation after OCU410 administration
Laboratory parameters including serum chemistry and hematology | 12 months (Screening to 12 months post OCU410 administration)
  Blood samples will be collected for the assessment to determine a change from baseline after OCU410 administration.

OTHER OUTCOMES:
Structural Outcome: Change Using Qualitative and quantitative assessments of autofluorescence pattern (FAF) | 12 months (Screening to 12 months post OCU410 administration)
  Changes in the intensity of FAF will be evaluated from the baseline measurements, to assess the loss of retinal layers.
Changes in National Eye Institute Visual Function Questionnaire 25 (NEI-VFQ25) | 12 months (Screening to 12 months post OCU410 administration)
  The National Eye Institute Visual Function Questionnaire 25 (NEI-VFQ25) questionnaires will be completed to assess the impact of vision on quality of subject's life.
Change From Baseline in Mean Threshold Sensitivity (MAIA) | 12 months (Screening to 12 months post OCU410 administration)
  Mean threshold sensitivity of all points will be determined to assess the macular functional response and determine GA progression.
Change from Baseline in drusen volume using SD-OCT | 12 months (Screening to 12 months post OCU410 administration)
  Measurement of change in drusen volume will be determined using Spectral Domain OCT measurements.
Change from Baseline in Exploratory Structural Imaging parameters including EZ and RPE loss | 12 months (Screening to 12 months post OCU410 administration)
  Measurement of change in structural parameters will be determined using imaging from Spectral Domain OCT measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Murthy Chavali, Ph.D, Study Director — Ocugen
Locations (12):
- United States (12):
  - Associated Retina Consultants, Phoenix, Arizona
  - Advanced Research, LLC, Coral Springs, Florida
  - Miidwest Eye Institute, Carmel, Indiana
  - Mississippi Retina Associates, Jackson, Mississippi
  - The Retina Institute, St Louis, Missouri
  - Mid Atlantic Retina, Cherry Hill, New Jersey
  - Duke Eye Center, Durham, North Carolina
  - The University of Pittsburgh, Pittsburgh, Pennsylvania
  - B) Retina Consultants of Texas, Bellaire, Texas
  - A) Retina Foundation of the Southwest, Dallas, Texas
  - Valley retina Institute, McAllen, Texas
  - Gundersen Health System, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No